CLINICAL TRIAL: NCT01530490
Title: Prevention of Ovarian Hyperstimulation Syndrome in GnRH Agonist IVF Cycles: Randomized Study Comparing Hydroxyethyl Starch Versus Cabergoline and Hydroxyethyl Starch
Brief Title: Cabergoline and Hydroxyethyl Starch in Ovarian Hyperstimulation Syndrome Prevention
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital de Cruces (Other)
Responsible Party: Principal Investigator, Roberto Matorras, Head of reproduction Unit, Hospital de Cruces
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIC0754
Record Dates: First submitted 2012-01-26; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Complications Associated With Artificial Fertilization; Disorder of Endocrine Ovary
Keywords: IVF; ovarian hyperstimulation syndrome; cabergoline; hydroxyethyl starch; prevention
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Cabergoline; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemoes (No Intervention)
- Cabergoline (Experimental): cabergoline
  Interventions: Drug: Cabergoline and Hydroxyethyl Starch; Drug: Hydroxyethyl Starch

INTERVENTIONS:
Drug: Cabergoline and Hydroxyethyl Starch — 0.5mg
  Other Names: Dostinex
  Arms: Cabergoline
Drug: Hydroxyethyl Starch — 0.5 mg cabergoline administration 8 days
  Other Names: Hemoes
  Arms: Cabergoline

SUMMARY:
The purpose of this study is to assess whether, in GnRH agonist in vitro fertilization (IVF) cycles, where there is a risk of ovarian hyperstimulation syndrome (OHSS), the addition of cabergoline to the hydroxyethyl starch infusion could decrease OHSS incidence and severity.

DETAILED DESCRIPTION:
Women undergoing IVF cycles with GnRH agonist protocols, at risk of OHSS (more than 20 follicles observed larger than 12 mm in diameter and/or estradiol levels of 3000-5000 pg/mL).

Slow infusion of 500 ml of 6% HES during follicular aspiration alone or combined with 0.5 mg cabergoline administration for 8 days, starting on the day of hCG administration.

ELIGIBILITY:
Inclusion Criteria:

* to be at risk of OHSS were invited to participate in the study

Exclusion Criteria:

* age > 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
risk of ovarian hyperstimulation syndrome | 12 days

SECONDARY OUTCOMES:
pregnancy rate | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Matorras, MD, PhD, Principal Investigator — Hospital Cruces

REFERENCES:
- [Derived] Matorras R, Andres M, Mendoza R, Prieto B, Pijoan JI, Exposito A. Prevention of ovarian hyperstimulation syndrome in GnRH agonist IVF cycles in moderate risk patients: randomized study comparing hydroxyethyl starch versus cabergoline and hydroxyethyl starch. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):439-43. doi: 10.1016/j.ejogrb.2013.07.010. Epub 2013 Aug 8. PMID 23932181